CLINICAL TRIAL: NCT06336200
Title: Kinesiophobia in Patients With Total Knee Arthroplasty
Brief Title: Knee Osteoarthritis and Kinesiophobia
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, Karabuk University
Other Study IDs: Karabuk-006
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Kinesiophobia
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Higher Kinesiophobia: It is a group with a high level of kinesiophobia according to the "Tampa kinesiophobia scale".
- Lower Kinesiophobia: It is a group with a low level of kinesiophobia according to the "Tampa kinesiophobia scale".

SUMMARY:
Kinesiophobia after total knee arthroplasty is an important parameter affecting recovery. However, the relationship between kinesiophobia and the factors it may cause is not clear. Therefore, this study aimed to examine the relationship between kinesiophobia, pain, fear of falling, mobility and proprioception in the early period after total knee arthroplasty.

DETAILED DESCRIPTION:
Various biopsychosocial factors affect the recovery process and quality of life after total knee arthroplasty. This situation reaches a level that can affect the daily life activities of patients, especially in the long term. Especially kinesiophobia is one of these factors. This condition also affects the proprioceptive sense in the knee, the capacity to move and the fear of falling. However, studies have generally examined long-term effects after total knee arthroplasty. Early studies are limited in number. More studies are needed to better understand the relationship between kinesiophobia and biopsychosocial factors. Additionally, the lack of relationship between the patients' kinesiophobia level, fear of falling, and proprioception in the early period after TKA draws attention. Therefore, this study aimed to examine the relationship between kinesiophobia, pain, fear of falling, mobility and proprioception in the early period after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-80
* Total knee arthroplasty surgery due to knee osteoarthritis
* Volunteering to participate in the study

Exclusion Criteria:

* Previously had knee surgery or fracture
* Diagnosed with rheumatoid arthritis
* Those with severe obesity (BMI > 40 kg/m2)
* Those with sensory and motor impairments
* Revision knee arthroplasty planned
* Venous thromboembolism
* Neurological diseases (MS, Parkinson, etc.)
* Early post-surgical complications

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who have undergone total knee arthroplasty surgery will be included in the study. Patients will be divided into two groups, high and low kinesiophobia levels, according to the Tampa Kinesiophobia Scale.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | Baseline
  Tampa Kinesiophobia Scale will be used to measure the level of fear of movement and re-injury. In this scale, a score ranges from 17 to 68, and an increase in the score means an increase in kinesiophobia. A score of 39.5 and above indicates the presence of high kinesiophobia.
Severity of pain | Baseline
  Visual analog scale (VAS) will be used to evaluate individuals' level of knee pain. A value of 0 indicates no pain, a value of 10 indicates very high pain.
Functional mobility | Baseline
  'Timed Up and Go Test' will be used to evaluate the mobility and functions of the patients.
Proprioception | Baseline
  Patients' knee joint proprioception sense will be measured with the 'Knee Joint Position Sense Test'. The angle of deviation from the target angle will be determined.
Fear of falling | Baseline
  While performing daily living activities, self-confidence and fear of falling will be evaluated with The Falls Efficacy Scale-International. A score between 16-65 is taken and as the total score increases, the probability of falling increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Pursaklar Public Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No